CLINICAL TRIAL: NCT06387225
Title: Early and Objective Assessment of Neurological Prognosis in Cardiac Arrest Patients
Acronym: HYPERION-2
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC23_0248
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Cardiac Arrest; Neurologic Symptoms; Intensive Care Neurological Disorder
MeSH Terms: conditions — Heart Arrest; Neurologic Manifestations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cerebral lesions are responsible for two thirds of deaths in patients admitted to intensive care following cardiac arrest. Patients with neurological lesions should be the priority target for neuroprotective interventions, which are the cornerstone of post-cardiac arrest care (allowing a reduction in the burden of care for patients without this type of lesion). Furthermore, these interventions must be based on a precise assessment of the severity of these brain lesions: carrying out neuro-protective interventions in patients without brain lesions exposes these patients to unnecessary treatment potentially associated with adverse effects without any possible benefit. However, the early assessment of neurological prognosis, particularly on admission to intensive care, is an area where there is little research and where it is not possible to obtain a precise and reproducible assessment. Several tools can be used to assess this prognosis at an early stage: anamnesis and characteristics of the cardiac arrest and the patient's comorbidities, imaging, electrophysiology and biomarkers.

To assess the predictive value of early biomarker testing in patients resuscitated after cardiac arrest, whatever the cause, the investigators plan to conduct a prospective observational multicentre trial.

It is important to bear in mind that the aim of this study is not to assess the long-term prognosis of patients suffering cardiac arrest in order to take measures to limit or discontinue active therapies, but simply to provide a reliable tool, simple and quick to use, in order to be able to identify a sub-population of patients who should be the subject of preferential neuro-protection measures, and conversely to simplify management (moderate temperature control, early cessation of sedation, early extubation) for patients with no neurological lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to intensive care with out-of-hospital cardiac arrest
* Comatose on admission (defined by a Glasgow score ≤ 8)
* Informed relative who has consented to the patient's participation in the study or inclusion under emergency procedure if the relative is absent at the time of inclusion

Exclusion Criteria:

* In-hospital cardiac arrest
* Age < 18 years
* Person under guardianship or legal protection
* Prior inclusion in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be included on admission to intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 608 (Estimated)
Dates: Start 2025-02-02 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Dosage of biomarker UCHL-1 (Ubiquitin carboxy-terminal hydrolase L1) at the time of admission to intensive care | at ICU admission
  Determine an assay threshold value admission to the intensive care unit to predict membership of a homogeneous group with favorable neurological outcome at D90
Dosage of biomarker GFAP (Glial fibrillary acidic protein) at the time of admission to intensive care | at ICU admission
  Determine an assay threshold value admission to the intensive care unit to predict membership of a homogeneous group with favorable neurological outcome at D90
Neurological outcome at D90 assessed by modified Rankin scale (mRS) | 90 days after patient enrolment in the study
  Determine an assay threshold value admission to the intensive care unit to predict membership of a homogeneous group with favorable neurological outcome at D90

SECONDARY OUTCOMES:
Dosage of biomarkers UCHL-1 ((Ubiquitin carboxy-terminal hydrolase L1) at the time of admission to intensive care | at ICU admission
  Determine prognostic value (positive and negative predictive value (PPV/NPV), positive and negative likelihood ratio (LR+/LR-) of each biomarker separately according to the threshold on admission.
  Determine the value of combining the two biomarkers at admission.
Dosage of biomarkers GFAP (Glial fibrillary acidic protein) at the time of admission to intensive care | at ICU admission
  Determine prognostic value (positive and negative predictive value (PPV/NPV), positive and negative likelihood ratio (LR+/LR-) of each biomarker separately according to the threshold on admission.
  Determine the value of combining the two biomarkers at admission.
Dosage of biomarkers UCHL-1 (Ubiquitin carboxy-terminal hydrolase L1) at 4 hours for recovery of effective cardiac activity (RACS) | at 4 hours for recovery of effective cardiac activity (RACS)
  Determine a threshold value at H4 for recovery of effective cardiac activity (RACS) to predict membership of a homogeneous group with a favorable neurological outcome at D90.
  Determine interest of combining the two biomarkers at H4 of the RACS.
Dosage of biomarkers GFAP( Glial fibrillary acidic protein) at 4 hours for recovery of effective cardiac activity (RACS) | at 4 hours for recovery of effective cardiac activity (RACS)
  Determine a threshold value at H4 for recovery of effective cardiac activity (RACS) to predict membership of a homogeneous group with a favorable neurological outcome at D90.
  Determine interest of combining the two biomarkers at H4 of the RACS.
Neurological outcome at D90 assessed by modified Rankin scale (mRS) ranging from 0 to 6 | 90 days after patient enrolment in the study
  Determine a threshold value at H4 for recovery of effective cardiac activity (RACS) to predict membership of a homogeneous group with a favorable neurological outcome at D90.
  A score of 0 to 3 is considered a favorable neurological outcome.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHD Vendée, La Roche-sur-Yon
  - CHU Nantes, Nantes
  - APHP - Hôpital Cochin, Paris
  - CH Saint-Nazaire, Saint-Nazaire